CLINICAL TRIAL: NCT02678052
Title: Organization of Teratology Information Specialists (OTIS) Vedolizumab Pregnancy Exposure Registry
Brief Title: OTIS Vedolizumab Pregnancy Exposure Registry
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: The Organization of Teratology Information Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5001; EUPAS11681 (Registry Identifier: ENCePP)
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Colitis, Ulcerative; Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: No Chronic Disease: Pregnant women without a current diagnosis of any chronic disease with no exposure to any biological agent and at any time from first day of last menstrual period (LMP) will be observed for up to 1 year.
- Cohort 2: UC/CD Prospective Cohort: Pregnant women with current diagnosis of UC or CD with exposure to Entyvio or other biologic agents during pregnancy at any dose, and at any time from first day of LMP will be observed for up to 1 year.
  Interventions: Drug: Vedolizumab; Biological: Other Biological Agent

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab exposure
  Other Names: Entyvio
  Groups: Cohort 2: UC/CD Prospective Cohort
Biological: Other Biological Agent — Other Biological Agent exposure
  Groups: Cohort 2: UC/CD Prospective Cohort

SUMMARY:
The purpose of this study is to assess the prevalence of major structural birth defects in infants of female participants with ulcerative colitis (UC) or Crohn's disease (CD) exposed to vedolizumab during pregnancy, compared to participants with UC or CD exposed to other biologic agents.

DETAILED DESCRIPTION:
The drug being observed in this study is called Vedolizumab. Vedolizumab is approved for the treatment of adult participants with moderately to severely active UC and CD who achieved an inadequate response, had a loss of response, or were intolerant to conventional and/or biologic treatments. This study will look at any possible association between vedolizumab and pregnancy outcome, including the health of the mother, fetus, and infant in the female with planned and unplanned pregnancies and who are at least 1 dose exposed at any time from last menstrual period (LMP) during pregnancy to vedolizumab (Entyvio) or other biological agents for UC or CD.

The study will enroll approximately 200 pregnant female participants drawn from 3 sources: OTIS Network, pregnant women who spontaneously contact the study research center or the sponsor or who are referred by their health care practitioners (HCP) in North America and women in North America who become pregnant while participating in other Entyvio clinical studies being undertaken by the sponsor. Participants will be assigned to one of the two cohorts:

* No chronic disease prospective cohort
* UC/CD prospective cohort All participants will be observed throughout the study. All participants will be asked to record all medications (including dose, frequency, and route), any additional exposures or events as the pregnancy progresses in a pregnancy diary.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 6 years. Cohort enrollment will be done before 20 weeks of gestation period and intake interviews would be scheduled telephonically. Schedule of intake interviews of participants will depends upon the duration of LMP prior to enrollment of participants in study. Outcome interview would be conducted within 0 to 6 weeks after delivery, dysmorphological examination of live infants would be conducted within 0 to 12 months after delivery and pediatric medical record review and questionnaire would be held 1 year after delivery.

ELIGIBILITY:
Inclusion Criteria:

For the UC/CD Prospective Cohort:

1. Is a currently pregnant woman with UC or CD,
2. Has exposure to Entyvio or other biologic agents at any dose, and at any time from first day of LMP,
3. Has enrolled no later than 19 completed weeks after LMP.
4. Agrees to the conditions and requirements of the study including the interview schedule, release of medical records, and the physical examination of live born infants.

   For the 'no chronic disease' Prospective Cohort:
5. Is a currently pregnant woman with no chronic disease.
6. Has no exposure to any biological agent and at any time from first day of LMP,
7. Has enrolled no later than 19 completed weeks after LMP.
8. Agrees to the conditions and requirements of the study including the interview schedule, release of medical records, and the physical examination of live born infants.

Exclusion Criteria:

For the UC/CD Prospective Cohort:

1. Is greater than (>) 19 completed weeks gestation prior to enrollment,
2. Has first contact with OTIS after prenatal diagnosis of any major structural defect,
3. Has enrolled in this registry with a previous pregnancy,
4. Has had an exposure to the known or suspected human teratogens: Chlorambucil. Cyclophosphamide, Mycophenylate mofetil.

   For the 'no chronic disease' Prospective Cohort:
5. Is >19 completed weeks gestation prior to enrollment,
6. Has first contact with OTIS after prenatal diagnosis of any major structural defect,
7. Has enrolled in this registry with a previous pregnancy,
8. Has had an exposure to the known or suspected human teratogens: Chlorambucil, Cyclophosphamide, Mycophenylate mofetil.

Note: women exposed to Entyvio during pregnancy but not meeting the above criteria can enroll into the Entyvio pregnancy exposure case series component of this registry.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant woman with or without UC or CD with exposure to Entyvio or any other biological agent (only for women with UC or CD) during pregnancy will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Major Structural Birth Defects Identified in Infants After Birth | Baseline up to 1 year
  A major structural defect is defined as a defect that has either cosmetic or functional significance to the child (eg, a cleft lip), as defined by the Centers for Disease Control and Prevention (CDC). These defects in aggregate typically occur in less than (<) 4% of the general population. Over 100 specific structural defects are considered to be major. Baseline will be considered as the time of birth of child.

SECONDARY OUTCOMES:
Minor Structural Birth Defects Identified in Infants After Birth | Baseline up to 1 year
  A minor structural defect is defined as a defect that has neither cosmetic nor functional significance to the child (for example: complete 2,3 syndactyly of the toes) and will be identified using a study-related checklist incorporated into the study dysmorphology examination of live born infants. Baseline will be considered at the time of birth of child.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda; Study Director, Study Director — The Organization of Teratology Information Specialists
Locations (1):
- San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b60394db2bf003ab4a249??page=1&idFilter=Vedolizumab-5001